CLINICAL TRIAL: NCT05830370
Title: Prevalence of Intestinal Parasitic Infections in Irritable Bowel Syndrome Patients in Sohag, Egypt
Brief Title: Prevalence of Intestinal Parasitic Infections in Patients With Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Mahmoud Ahmed, Demonstrator at medical parasitology department., Sohag University
Other Study IDs: Soh-Med-23-04-23MS
Record Dates: First submitted 2023-04-12; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; entamoeba; histolytica; Blastocystis; hominis; chronic abdominal pain; diarrhea; defecation; constipation; bloating; Trichinella; Cryptosporidium
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — stool specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: patients complaining of symptoms of IBS fulfilling the Rome criteria , such as abdominal discomfort, diarrhea, and constipation, bloating with any age & sex groups from different locations.
- control: healthy individuals not suffering from IBS symptoms such as abdominal discomfort, diarrhea, and constipation, bloating.

SUMMARY:
Irritable bowel syndrome (IBS) is common medical disorder and represent a group of diseases of the gastrointestinal tract that is characterized by chronic abdominal pain , bloating , passage of mucus or straining with bowel movements, sense of incomplete evacuation after bowel movements or sense of urgency to move the bowels.Several parasites including Entamoeba. histolytica, Giardia spp., Blastocystis. hominis, and Trichinella spp. have been discussed as contributing factors to the development of IBS.

B. hominis is one of the most common human intestinal protozoa in both developing and developed countries. some studies have reported a significant association between the parasitic infections, especially Blastocystis, and IBS.Cryptosporidium has been reported in IBS patients, with the onset of gastrointestinal symptoms after an acute episode of cryptosporidiosis despite recovery and parasite clearance.Numerous studies have been conducted to evaluate the association between the parasitic infections and IBS.

Aim of the work:

To detect prevalence of intestinal parasitic infections in irritable bowel syndrome patients in sohag.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of symptoms of IBS, such as abdominal discomfort, diarrhea, and constipation, bloating with any age & sex groups

Exclusion Criteria:

* Patients have celiac disease, gastrointestinal malignancies , inflammatory bowel disease , HIV , and those on immunosuppression and those who had been recently taking antibiotics within the previous four weeks and anti-parasitic drugs within the previous two weeks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: samples will be collected from outpatients complaining of symptoms of IBS fulfilling the Rome criteria , such as abdominal discomfort, diarrhea, and constipation, bloating with any age & sex groups from different locations (cities and village).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
To detect prevalence of intestinal parasitic infections in irritable bowel syndrome patients in sohag. | 16 weeks following the startpoint of the study.
  will collect 200 stool samples : 100 samples will be collected from patients complaining of symptoms of IBS fulfilling the Rome criteria , such as abdominal discomfort, diarrhea, and constipation, bloating with any age & sex groups from different locations (cities and village) And 100 samples healthy controls.the samples will be examined for parasitological examination to detect prevalence of intestinal parasitic infections in irritable bowel syndrome patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided